CLINICAL TRIAL: NCT03676530
Title: Pain Reduction in Tibial Stress Syndrome Using Compression Garments
Brief Title: Pain Reduction in Tibial Stress Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Marion V. Sanders, Principal Investigator, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TSS2018
Record Dates: First submitted 2018-08-16; First posted 2018-09-18 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Tibial Stress Syndrome

STUDY DESIGN:
Intervention Model Description: Pro-Tec Shin Splints Compression Wrap
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relative Rest (Control) (No Intervention): Male/Female Military Trainees with symptoms consistent with Tibial Stress Syndrome. No compression. Standard of care therapy includes relative extremity rest, stretches and graduated run program.
- Compression Garments (Experimental): Male/Female Military Trainees with symptoms consistent with Tibial Stress Syndrome. Standard of care therapy includes compression garments worn, stretches and graduated run program.
  Interventions: Device: Pro-Tec Shin Splint Compression Wrap

INTERVENTIONS:
Device: Pro-Tec Shin Splint Compression Wrap — EVA Foam pad compression device with Velcro straps that is placed over tibial site of pain.
  Arms: Compression Garments

SUMMARY:
This study is intended to determine if compression garments effectively reduce pain in the treatment of tibial stress syndrome (TSS) in the military population. The study will include diagnoses of shin splints, which is medically known as tibial stress syndrome and medial tibial stress syndrome, and compare a treatment group using compression garments to a control group using passive recovery. Both groups will engage in a progressive walk-to-run program. The outcomes will be measured by comparison in pain scales pre and post treatments. The ability to perform a two mile run without pain symptoms will be assessed at the conclusion of the study by participant's self-reported evaluation. The TSS screening questionnaire will be obtained at each medical encounter to include the initial visit and follow-up visits at the four and eight week (+/- 3 days) marks. The self-reported 2-mile run evaluation is included on the TSSS questionnaire.

DETAILED DESCRIPTION:
The study objective is to determine whether use of compression garments in the treatment of tibial stress syndrome will reduce pain compared with passive recovery alone.

Specific aims include evaluation of Visual Analog Scale (VAS) when utilizing compression garments and passive recovery and a self-reported pain free running assessment by the participant. VAS evaluation will occur at initial encounter, four weeks from treatment initiation, and then again at eight weeks from treatment start. The follow up time frames will have a ± three days to allow flexibility of the participant to follow up. The study will be assessed with a 60 day evaluation period to coincide with previous study time periods as well as the ability to lessen the possibility of participants lost to follow up that may be relocated due to military orders. Assessment of functionality, symptomatic criteria, and determination if further care is required will occur at each visit. A self-reported pain free running assessment will be collected via questionnaire at the conclusion of the study.

The investigators intend to prove that compression garments will better reduce pain symptoms in the treatment of tibial stress syndrome (shin splints) compared with passive recovery alone.

Conduct a prospective randomized control trial with the objective of determining if the application of compression garments for the symptomatic treatment of tibial stress syndrome produces improved rates of pain relief and activity tolerance compared to the control of passive recovery.

Subject population will be gathered from Fort Sam Houston McWethy TMC patients who consist of active duty trainees for all military branches of service. Male and female participants from 18-45 years of age presenting with leg pain consistent with tibial stress syndrome will be considered for this study. Age limitation is based on assumed increase in potential confounders related to previous injury or pre-existing musculoskeletal conditions. Approximately 42 participants are required based on comparison with previous studies. This includes a 20 percent addition to account for participants lost to follow-up. Control group will be treated with passive recovery only.

ADHOC report on international classification of diseases tenth revision, clinical modification (ICD10) will be obtained for local comparisons of lower extremity diagnoses.

The inclusion criteria consist of:

* Patients of the McWethy TMC
* Able to provide informed consent (of sound mind)
* Acute or acute on chronic musculoskeletal pain of lower extremity
* 18-45 years of age
* Active duty military trainees of all service branches assigned to unit on Ft Sam Houston
* Pain at presentation indicated on Visual Analog Scale (VAS). All scores indicated on the VAS will be accepted.

The exclusion criteria consist of:

* Patients outside of the McWethy TMC or not assigned to a unit on Ft Sam Houston
* Patient with lower extremity pain not consistent with tibial stress syndrome
* Participants with open wounds of the lower extremity
* Temperature greater than 38˚ Celsius (100.4 Fahrenheit)
* Pain associated with current diseases (neurologic/rheumatologic/cancer)
* Active infection at injury location
* Patients younger than 18 or older than 45 years of age

This research will be a prospective, randomized control trial. Subjects will be randomly assigned to one of two conditions: use of compression garments (CG) in the treatment group or passive recovery in the control group. Subjects will be randomized to either the treatment or the control group through use of an envelope with separate cards indicating either "relative rest" or "compression garment" on each individual card within the envelope. The envelope will be maintained by the PI and/or AI associated with this study. The card within the envelope will be selected by the study participant at the initial visit after the physical examination has been completed.

Active duty Service members in training status arriving to the McWethy TMC with acute or acute on chronic shin pain as a chief complaint will be considered for the study. Only those meeting the inclusion criteria will be invited to take part in this study. Participants enrolled in the study will be randomized to either control (n=21) or CG (n=21) groups.

Each subject will be placed on a no run or walk profile for 60 days with the caveat of gradual return to run expected. The graduated walk-to-run progression program will be in accordance with Lackland Air Force Base Physical Therapy protocols. Subjects randomized to the passive recovery (control) group will follow two weeks of total lower extremity rest, excluding normal daily activities, while gradually integrating impact activity tolerance to running over the remaining six weeks of the study. Subjects randomized to the CG group will be measured for orthotics in accordance with manufacturer's recommendations and instructed on the proper wear and use during their initial visit with the provider. CG will be worn at rest for the initial two weeks following the initial encounter and then with activity between weeks two and eight ± three days. CG may be used unilaterally or bilaterally depending on the chief complaint of the subject. The subject will be instructed to continue wear of the CG for the duration of the recommended treatment timeline unless an individual's pain scale of 0 has been achieved and maintained throughout the study time period. The participant will continue wear of the compression garment throughout the day for the first two weeks and then with activity for the next six weeks. If the participant develops any worsening of lower extremity symptoms they will be advised to discontinue use and follow up with their primary care provider. This data will be included into the research.

Each subject who consents to participate in the current study will complete a study-specific questionnaire to obtain demographic information such as gender, age, and branch of service. Demographic information will be collected for follow-up access and ensure contact with each participating member is included. This information will be used for the purpose of follow-up or research contact only. No PHI will be included in the data analysis or into research documentation for any other purpose and will not be included in the final documentation or research findings annotation. Additionally, information regarding number of days per week each subject runs will be collected. Specifics on their perceived shin pain will be ascertained that incorporates location, pain with ambulation, pain with running, pain with sports activity, unilateral or bilateral symptom complaints, and pain at rest.

Furthermore, provider questioning and physical exam will include appearance of foot arch at standing, roll of foot with ambulation, tenderness on palpation, pain with provocative tests, pertinent historical evidence, range of motion, and body mass index. The diagnosis of tibial stress syndrome will rely on clinical examination only. The diagnosis of medial tibial stress syndrome has been condensed to tibial stress syndrome to ensure that a broader range of tibial pain is included. Two common sites of exercise-induced tibial pain have been described, posteromedial and more proximally anterolateral which reflects the posterior and anterior tibial compartments, respectively.

CG in the treatment of TSS pain is likely to be a simple intervention that utilizes a patient-centered strategy to elicit both short-term and long-term therapeutic benefits. Knowledge of the range, individuality, and varied temporal patterns of treatment outcomes can guide potential patients, clinicians, health care providers, and researchers. An informed characterization of the treatment process in any intervention is needed to support appropriate care and optimal results. Performing a nested qualitative study within the pragmatic clinical trial will provide depth and meaning to the health-related outcome measures. Each participant will be screened using a satisfaction questionnaire after the treatment phase to obtain an account of his or her receiving the specific treatment related to shin splint pain in the McWethy TMC.

The primary outcome measure will be determined by using the visual analog scale (VAS) at rest and compared to with impact activities such as running. VAS is a unidimensional pain intensity scale; a 10-cm (100-mm) line on which the subject is asked to place a mark that corresponds with his or her current pain intensity. The secondary outcomes are, pain time-response after treatment, performance using subjective activity data collection, and satisfaction using a binomial (yes/no), and the need for further evaluation after study completion, which will be obtained during follow up at the four week timeframe or via phone follow-up if member is unable to schedule a face to face visit.

The primary outcome measure (pain level, assessed using the VAS) will be collected at baseline, four weeks (+/- 3 days), and eight weeks (+/- 3 days) after the initial encounter. The secondary outcomes (time-response, performance and functionality, satisfaction) will be measured at baseline, four weeks post initial encounter (+/- 3 days), and eight weeks (+/- 3 days) post initial encounter. Additional data collected, such as pain at rest and with activity, and physical examination findings will be obtained during the medical visits and used into data collection.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the McWethy TMC
* Able to provide informed consent (of sound mind)
* Acute or acute on chronic musculoskeletal pain of lower extremity
* 18-45 years of age
* Active duty military trainees of all service branches assigned to unit on Ft Sam Houston
* Pain at presentation indicated on Visual Analog Scale (VAS). All scores indicated on the VAS will be accepted

Exclusion Criteria:

* Patients outside of the McWethy TMC or not assigned to a unit on Ft Sam Houston
* Patient with lower extremity pain not consistent with tibial stress syndrome
* Participants with open wounds of the lower extremity
* Temperature greater than 38˚ Celsius (100.4 Fahrenheit)
* Pain associated with current diseases (neurologic/rheumatologic/cancer)
* Active infection at injury location
* Patients younger than 18 or older than 45 years of age

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in reported pain scores using compression garments | Initial visit, 4 week follow up, 8 week follow up
  scored against Visual Analog Pain Scale from 0 to 100 millimeters with 0 being no pain and 100 being the worst pain possible

CONTACTS AND LOCATIONS:
Locations (1):
- SAMMC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Possible publication.